CLINICAL TRIAL: NCT06555614
Title: Prospective and Retrospective, Single Center, Case-control, Investigator-initiated, Observational Study to Evaluate the Safety of Acellular Dermal Matrix Processed by the Supercritical CO2 Technology in Breast Reconstruction With Implants
Brief Title: Evaluation of Safety of Acellular Dermal Matrix(ADM) in Breast Reconstruction
Acronym: ADM
Status: Recruiting | Type: Observational
Sponsor: DOF Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-01-005
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer Female; Breast Reconstruction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test Group: A prospectively selected group that will receive breast reconstruction surgery with an acellular dermal matrix called "SC Derm Recon," which is processed using carbon dioxide supercritical fluid technology.
  Interventions: Other: Acellular Dermal Matrix(ADM)
- Control Group: A retrospectively selected group that has undergone breast reconstruction surgery with an acellular dermal matrix processed using chemical detergents.
  Interventions: Other: Acellular Dermal Matrix(ADM)

INTERVENTIONS:
Other: Acellular Dermal Matrix(ADM) — A comparison of the short-term complications associated with acellular dermal matrix in the test group and the control group.

SUMMARY:
The goal of this observational study is to evaluate the safety of Acellular Dermal Matrix(ADM) processed by CO2 supercritical fluid technology against other acellular dermal matrix products from different companies that have been washed with detergents in patients undergoing breast reconstruction surgery with implants due to the breast cancer.

DETAILED DESCRIPTION:
Outline:

The total number of study subjects is 120, with 60 people recruited prospectively into the test group and 60 people retrospectively into the control group.

The test group will receive SC Derm Recon(ADM processed by CO2 supercritical fluid technology) during the implant-based breast reconstruction surgery.

The control group will be retrospectively and consecutively selected from medical records of patients who underwent implant breast reconstruction using ADM from other companies between March 1, 2021, and March 31, 2024.

After surgery, patients will be followed up at 2 weeks, 4 weeks, and 12 weeks.

Primary Objectives

I. To assess whether the test group with applying the ADM processed by the supercritical fluid technology will have less short-term major complications than the control group with the ADM processed by detergents.

ELIGIBILITY:
Inclusion Criteria:

1. Prospective subjects (Test group) 1) Adult women aged 19 to 79 years. 2) Patients who received SC DERM® Recon, an acellular dermal matrix product, during breast reconstruction surgery with implants following a mastectomy due to breast cancer. 3) Individuals who have voluntarily provided written informed consent after receiving an explanation of the study's purpose and methods, are willing to comply with the study protocol, and are willing to visit the hospital for the evaluation of observational parameters.
2. Retrospective Medical Record Collection 1) Patients who received an acellular dermal matrix product during breast reconstruction surgery with implants following a mastectomy due to breast cancer at Seoul National University Hospital between March 1, 2021, and March 31, 2024.

Exclusion Criteria:

1. Prospective subjects (Test group) 1) Individuals deemed inappropriate for study participation by the principal investigator or other investigator's judgement. (e.g., those unable to undergo the required tests for this study).
2. Retrospective Medical Record Collection 1) Patients who received an acellular dermal matrix product but have no recorded follow-up visits after application.

Ages: 19 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female Patients who received an acellular dermal matrix during breast reconstruction surgery with implants following a mastectomy due to breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence Rate(%) of Major Short-Term Complications Over 12 Weeks Post-Application of ADM | From the day of operation of breast reconstruction to 12weeks
  The primary endpoint is to compare and evaluate the incidence rate(%) of major short-term complications over 12 weeks following the application of acellular dermal matrix (ADM).

CONTACTS AND LOCATIONS:
Overall Officials: Kiyong Hong, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: National Health Insurance: Early Treatment Increases Survival Rates for Breast Cancer Patients, with a 6.9% Increase Over the Past 5 Years. Press Release, 2023-05-26. — https://www.akomnews.com/bbs/board.php?bo_table=news&wr_id=53470
- See also: Disa JJ, McCarthy CM, Mehrara BJ, Pusic AL, Hu QY, Cordeiro PG. Postmastectomy reconstruction: an approach to patient selection. Plast Reconstr Surg. 2009 Jul;124(1):43-52. — https://pubmed.ncbi.nlm.nih.gov/19346999/
- See also: Colwell AS, Taylor EM. Recent Advances in Implant-Based Breast Reconstruction. Plast Reconstr Surg. 2020 Feb;145(2):421e-432e. — https://pubmed.ncbi.nlm.nih.gov/31985660/
- See also: Sigurdson L, Lalonde DH. MOC-PSSM CME article: Breast reconstruction. Plast Reconstr Surg. 2008 Jan;121(1 Suppl):1-12. — https://pubmed.ncbi.nlm.nih.gov/18182962/
- See also: Gabriel A, Maxwell GP. Discussion: Prepectoral Breast Reconstruction: A Safe Alternative to Submuscular Prosthetic Reconstruction following Nipple-Sparing Mastectomy. Plast Reconstr Surg. 2017 Sep;140(3):444-446. — https://pubmed.ncbi.nlm.nih.gov/28841598/
- See also: Sbitany H, Piper M, Lentz R. Prepectoral Breast Reconstruction: A Safe Alternative to Submuscular Prosthetic Reconstruction following Nipple-Sparing Mastectomy. Plast Reconstr Surg. 2017 Sep;140(3):432-443. — https://pubmed.ncbi.nlm.nih.gov/28574950/
- See also: Breuing KH, Warren SM. Immediate bilateral breast reconstruction with implants and inferolateral AlloDerm slings. Ann Plast Surg. 2005 Sep;55(3):232-9. — https://pubmed.ncbi.nlm.nih.gov/16106158/
- See also: Gamboa-Bobadilla GM. Implant breast reconstruction using acellular dermal matrix. Ann Plast Surg. 2006 Jan;56(1):22-5. — https://pubmed.ncbi.nlm.nih.gov/16374090/
- See also: Bindingnavele V, Gaon M, Ota KS, Kulber DA, Lee DJ. Use of acellular cadaveric dermis and tissue expansion in postmastectomy breast reconstruction. J Plast Reconstr Aesthet Surg. 2007;60(11):1214 — https://pubmed.ncbi.nlm.nih.gov/17459797/
- See also: Zienowicz RJ, Karacaoglu E. Implant-based breast reconstruction with allograft. Plast Reconstr Surg. 2007 Aug;120(2):373-81. — https://pubmed.ncbi.nlm.nih.gov/17632337/
- See also: Salzberg CA. Nonexpansive immediate breast reconstruction using human acellular tissue matrix graft (AlloDerm). Ann Plast Surg. 2006 Jul;57(1):1-5. — https://pubmed.ncbi.nlm.nih.gov/16799299/
- See also: Breuing KH, Colwell AS. Inferolateral AlloDerm hammock for implant coverage in breast reconstruction. Ann Plast Surg. 2007 Sep;59(3):250-5. — https://pubmed.ncbi.nlm.nih.gov/17721209/
- See also: Spear SL, Parikh PM, Reisin E, Menon NG. Acellular dermis-assisted breast reconstruction. Aesthetic Plast Surg. 2008 May;32(3):418-25. — https://pubmed.ncbi.nlm.nih.gov/18338102/
- See also: Preminger BA, McCarthy CM, Hu QY, Mehrara BJ, Disa JJ. The influence of AlloDerm on expander dynamics and complications in the setting of immediate tissue expander/implant reconstruction: a matched-cohort study. Ann Plast Surg. 2008 May;60(5):510-3. — https://pubmed.ncbi.nlm.nih.gov/18434824/
- See also: Ho G, Nguyen TJ, Shahabi A, Hwang BH, Chan LS, Wong AK. A systematic review and meta-analysis of complications associated with acellular dermal matrix-assisted breast reconstruction. Ann Plast Surg. 2012 Apr;68(4):346-56. — https://pubmed.ncbi.nlm.nih.gov/22421476/
- See also: Vidya R, Cawthorn SJ. Muscle-Sparing ADM-Assisted Breast Reconstruction Technique Using Complete Breast Implant Coverage: A Dual-Institute UK-Based Experience. Breast Care (Basel). 2017 Sep;12(4):251-254. — https://pubmed.ncbi.nlm.nih.gov/29070989/
- See also: Vidya R, Iqbal FM. A Guide to Prepectoral Breast Reconstruction: A New Dimension to Implant-based Breast Reconstruction. Clin Breast Cancer. 2017 Jul;17(4):266-271. — https://pubmed.ncbi.nlm.nih.gov/28190760/
- See also: Sigalove S, Maxwell GP, Sigalove NM, Storm-Dickerson TL, Pope N, Rice J, Gabriel A. Prepectoral Implant-Based Breast Reconstruction: Rationale, Indications, and Preliminary Results. Plast Reconstr Surg. 2017 Feb;139(2):287-294. — https://pubmed.ncbi.nlm.nih.gov/28121858/
- See also: Cattelani L et. al., One-Step Prepectoral Breast Reconstruction With Dermal Matrix-Covered Implant Compared to Submuscular Implantation: Functional and Cost Evaluation. Clin Breast Cancer. Clin Breast Cancer. 2018 Aug;18(4):e703-e711. — https://pubmed.ncbi.nlm.nih.gov/29275104/
- See also: Walter RJ, Matsuda T, Reyes HM, Walter JM, Hanumadass M. Characterization of acellular dermal matrices (ADMs) prepared by two different methods. Burns. 1998 Mar;24(2):104-13. — https://pubmed.ncbi.nlm.nih.gov/9625233/
- See also: Wainwright DJ. Use of an acellular allograft dermal matrix (AlloDerm) in the management of full-thickness burns. Burns. 1995 Jun;21(4):243-8. — https://pubmed.ncbi.nlm.nih.gov/7662122/
- See also: Lemer ML, Chaikin DC, Blaivas JG. Tissue strength analysis of autologous and cadaveric allografts for the pubovaginal sling. Neurourol Urodyn. 1999;18(5):497-503. — https://pubmed.ncbi.nlm.nih.gov/10494122/
- See also: Romo T 3rd, Sclafani AP, Sabini P. Reconstruction of the major saddle nose deformity using composite allo-implants. Facial Plast Surg. 1998;14(2):151-7. — https://pubmed.ncbi.nlm.nih.gov/11816205/
- See also: Neishabouri A, Soltani Khaboushan A, Daghigh F, Kajbafzadeh AM, Majidi Zolbin M. Decellularization in Tissue Engineering and Regenerative Medicine: Evaluation, Modification, and Application Methods. Front Bioeng Biotechnol. 2022 Apr 25;10:805299. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9081537/
- See also: Giang NN, Trinh XT, Han J, Chien PN, Lee J, Noh SR, Shin Y, Nam SY, Heo CY. Effective decellularization of human skin tissue for regenerative medicine by supercritical carbon dioxide technique. J Tissue Eng Regen Med. 2022 Dec;16(12):1196-1207. — https://pubmed.ncbi.nlm.nih.gov/36346009/